## PARTICIPANT CONSENT FORM KANSAS STATE UNIVERSITY

PROJECT TITLE: Stand Up Kansas: An intervention to reduce sedentary behavior in the workplace

APPROVAL DATE OF PROJECT: 09/18/2020 EXPIRATION DATE OF PROJECT: 07/06/2021

**LENGTH OF STUDY:** Approximately six months

PRINCIPAL INVESTIGATOR: Emily Mailey

## CONTACT NAME AND PHONE FOR ANY PROBLEMS/QUESTIONS:

Emily Mailey, emailey@ksu.edu, 847-224-1199

## IRB CHAIR CONTACT/PHONE INFORMATION:

If you have any questions about your rights as a research participant please contact the Kansas State University Institutional Review Board:

- Rick Scheidt, Chair, Committee on Research Involving Human Subjects, 203 Fairchild Hall, Kansas State University, Manhattan, KS 66506, (785) 532-3224.
- Cheryl Doerr, Associate Vice President for Research Compliance, 203 Fairchild Hall, Kansas State University, Manhattan, KS 66506, (785) 532-3224.

SPONSOR OF PROJECT: College of Health and Human Sciences, Kansas State University

**PURPOSE OF THE RESEARCH:** The overall purpose of this study is to evaluate the effectiveness of a program designed to help Kansas employees reduce their sitting time while working from home.

**PROCEDURES OR METHODS TO BE USED:** At the beginning of the study you will be asked to complete all of the assessments described below. Once we have collected all baseline data, you will be randomly assigned to one of four conditions: desk only, support program only, desk+support program, or waitlist control. If you are assigned to the desk only or desk+support condition, you will be asked to pick up a free height-adjustable desk on campus following your baseline assessments. If you are assigned to the support program or waitlist control condition, you will receive your height-adjustable desk after the post-program assessments (approximately four months later). The support program will consist of two individual coaching sessions, delivered virtually, and access to a variety of resources to help you sit less and move more in your home work environment.

All participants will repeat all of the assessments at the end of the 12-week intervention period, and again 12 weeks later.

## ASSESSMENTS:

All participants will complete the following tests and procedures in our laboratory (Lafene 3<sup>rd</sup> floor):

- *Metabolic blood panel*. Blood will be drawn from a quick finger stick to assess total cholesterol and fasting blood glucose.
- Body measurements. A trained research assistant will measure your height, weight, and waist circumference.
- *Blood pressure*. A trained research assistant will measure your blood pressure using an automated blood pressure cuff.

In addition, participants will complete the following assessments:

- *Questionnaires*: You will be asked to complete a series of questionnaires online. This should take about 10-15 minutes.
- Activity monitor: You may be asked to wear a motion sensor called an ActivPAL for 7 days at each time point (pending device availability). This small activity monitor is attached to your thigh and worn 24 hours per day during the wear period.

**RISKS OR DISCOMFORTS ANTICIPATED:** By increasing your time standing and moving during the workday, there is a chance of incurring minor injury and discomfort due to the intensified use of major muscle groups. To minimize muscle soreness we will recommend gradual increases in standing and/or light intensity activity in small, manageable bouts. Additionally, you may experience some discomfort with the fingerstick procedure. We will adhere to approved procedures to mitigate risk of COVID-19 infection, including staff/participant screenings prior to testing appointments, and requiring masks at all times during appointments.

**BENEFITS ANTICIPATED:** This study may or may not benefit you directly. Previous research has shown that reductions in sedentary behavior are associated with improvements in physical and mental health outcomes. Additionally, we hope the information gained from this study will contribute to the development of future programs to reduce sedentary behavior among employees.

**EXTENT OF CONFIDENTIALITY:** Confidentiality is assured for all participants with regard to any responses and information you provide. Your name or personal information will not be tied to any of your data, and your employer will not have access to your individual data. Your data will be coded with a study ID number that is linked to a participant list, and this list will be kept separate from study data. All participant information will be stored in a locked file cabinet that can only be accessed by approved research personnel. Your personal information may be given out only if required by law. If information from this study is published or presented at scientific meetings, your name and other personal information will not be used.

**IS COMPENSATION OR MEDICAL TREATMENT AVAILABLE IF INJURY OCCURS:** Kansas State University does not provide medical or hospitalization insurance coverage for participants in this research study nor will Kansas State University provide compensation for any injury sustained as a result of participation in this research study, except as required by law.

TERMS OF PARTICIPATION: I understand this project is research, and that my participation is completely voluntary. I also understand that if I decide to participate in this study, I may withdraw my consent at any time, and stop participating at any time without explanation, penalty, or loss of benefits, or academic standing to which I may otherwise be entitled.

I verify that my signature below indicates that I have read and understand this consent form, and willingly agree to participate in this study under the terms described, and that my signature acknowledges that I have received a signed and dated copy of this consent form.

| Participant Name: | |
|---------------------------------------|-------|
| Participant Signature: | Date: |
| Witness to Signature: (project staff) | Date: |